CLINICAL TRIAL: NCT01582867
Title: Studio Cross-Over Controllato Randomizzato Sul Dispositivo ArTis Con Hemocontrol in Emodiafiltrazione - SOCRATHE
Brief Title: HemoControl System Activated in Hemodiafiltration Treatments
Acronym: SOCRATHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Dasco S.p.A. (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1495
Record Dates: First submitted 2012-04-16; First posted 2012-04-23 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Renal Failure
Keywords: Hemodiafiltration; Hemodialysis; Sodium; Artis; renal failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HD and HDF (Experimental): During one part of the study (study phase A) patients will undergo hemodialysis (HD) treatments with Hemoscan over 2 weeks (Run-In period), followed by 12 HD sessions with HemoControl during the following 4 to 6 weeks. Separated by a one week wash out period, the same patients will be switched to On-Line Hemodiafiltration (HDF) treatments (study phase B), for a Run-In period of 2 weeks with Hemoscan, followed by 12 On-Line HDF sessions with HemoControl over the last 4 to 6 weeks of the study period.
  Interventions: Device: ARTIS hemodialysis system
- HDF and HD (Experimental): patients will be treated vice versa, starting with On-Line Hemodiafiltration (HDF) followed by hemodialysis (HD) with the same respective Run-In periods and a washout period as patients in Arm hemodialysis (HD) and Hemodiafiltration (HDF) .
  Interventions: Device: ARTIS hemodialysis system

INTERVENTIONS:
Device: ARTIS hemodialysis system — Software versions:
  Control Product: 8.06.01KA. Study Product: 8.06.01B_HC01
  Other Names: Artis™ hemodialysis system; HEMOCONTROL™; GAMBRO

SUMMARY:
The current study aims to assess the HemoControl prescription in On-Line Hemodiafiltration treatment.

DETAILED DESCRIPTION:
Hemodiafiltration (HDF) is a dialysis technique that allows the removal of high molecular weight toxic solutes exploiting the convective transport through the dialyzer membrane: at the same time, the HDF has a positive impact on the systemic hemodynamic, ameliorating in this way the tolerance of the treatment. Unfortunately, also the HDF therapy can be not well tolerated, introducing in the patients serious hypovolemia during the removal of the body water accumulated in the interdialytic period.

The HemoControl system, automatically controlling the relative blood volume change of the patient, avoids the onset of the hypovolemia. Today the HemoControl system can be used only during conventional hemodialysis treatments; the objective of this study is to combine the advantages of the intradialytic hemodynamic stabilization achievable by means of HemoControl with the inherent advantages, both of depurative and cardiovascular kind, typical of the Hemodiafiltration technique.

ELIGIBILITY:
Inclusion Criteria:

* A subject must meet ALL of the following inclusion criteria in order to participate in this study:

  * ESRD in chronic dialysis treatments for at least 3 months
  * Age ≥ 18 years
  * Body weight ≥ 40 kg
  * Blood flow rate ≥ 250 ml/min with a recirculation of the vascular access < 5%
  * Use of not fractioned heparin in continuous infusion as anticoagulant
  * Stable anticoagulation dosage over the last 6 treatments
  * Stable dialysis prescription (Qb, Qd, treatment time) over the last 6 treatments
  * Informed consent for participating to the study
  * Stable Haemoglobin concentration at beginning of the treatment lower than or equal to 14 g/dl.

Exclusion Criteria:

* A subject shall NOT participate in the study if he/she meets ANY of the following criteria:

  * HIV positivity
  * Active Hepatitis A, B or C
  * Pregnancy
  * Participating in other clinical investigations during the course of this study
  * Failed to release consent
  * Known coagulation disorders (clotting problems)
  * Known bleeding risk
  * Clinical or laboratory diagnosis of acute infection
  * Recent (last 4 weeks) surgical intervention
  * Therapy prescribed is only HD, HF or isolated UF mode
  * Active phase cancer,
  * Active phase immune disease.
  * Serious hemostasis disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Sodium mass balance | during dialysis treatment within 18 weeks
  * to determine whether the same HemoControl prescription is usable in On-Line Hemodiafiltration (HDF) and hemodialysis (HD) treatments and, if not,
  * to assess the existence of a proper HemoControl prescription in On-Line Hemodiafiltration (HDF) treatment.

SECONDARY OUTCOMES:
blood pressure | Pre-dialytic within 18 weeks
  difference between the pre-treatment systolic and diastolic blood pressures in On-Line Hemodiafiltration (HDF) and hemodialysis (HD) with respect to the control treatments
thirst perception | during dialysis within 18 weeks
  Average difference between the thirst score reported by the patient during On-Line Hemodiafiltration (HDF) and hemodialysis (HD) treatments with respect to the score reported during the control treatments
weight gain | between dialysis treatments within 18 weeks
  difference between the interdialytic weight gain in On-Line Hemodiafiltration (HDF) and hemodialysis (HD) treatments with respect to the control treatment

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Santoro, Dr., Principal Investigator — POLICLINICO SANT'ORSOLA MALPIGHI
Locations (1):
- Policlinico Sant'Orsola Malpighi, Bologna, (BO), Italy